CLINICAL TRIAL: NCT01408186
Title: Histamine-2 Receptor Antagonist Versus Proton-Pump Inhibitor for the Prevention of Recurrent Upper Gastrointestinal Bleeding (UGI) in High-risk Users of Low-dose Aspirin (ASA)
Brief Title: ASP (PPI_H2RA) Study-H2RA Versus PPI for the Prevention of Recurrent UGIB in High-risk Users of Low-dose ASA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APH Study
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: aspirin; PPI; H2RA
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Rabeprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rabeprazole (Active Comparator): Tablet 20mg daily for 12 months
  Interventions: Drug: Rabeprazole
- Famotidine (Active Comparator): Tablet 40mg daily for 12 months
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole 20 mg daily
  Other Names: Pariet
  Arms: Rabeprazole
Drug: Famotidine — Famotidine 40mg daily
  Other Names: Pepcidine
  Arms: Famotidine

SUMMARY:
Peptic ulcer bleeding associated with ASA or NSAIDs is a major cause of hospitalization in Hong Kong. The investigators previously showed that ASA or NSAIDs accounted for about half of all cases of hospitalizations for peptic ulcer bleeding. Currently, ASA use has contributed to about one-third of the bleeding ulcers admitted to the investigators hospital that serves a local population of 1.5 million.

In patients with acute coronary syndrome or acute ischemic stroke who develop ASA-induced bleeding peptic ulcers, whether ASA should be discontinued before ulcers have healed is a major dilemma. In another double-blind randomized trial, the investigators have shown that discontinuation of ASA after endoscopic treatment of bleeding ulcers was associated with a significantly increased in mortality within 8 weeks.

In the absence of safer aspirins, co-therapy with a gastroprotective drug remains the dominant preventive strategy. Given the vast number of people taking ASA, however, it is only cost-effective to identify and treat those who are at high risk of ulcer bleeding and who have a strong indication for ASA use. Data from observational studies and randomized trials have consistently shown that PPIs are effective in reducing the risk of ulcer bleeding associated with ASA. Other potential preventive strategies include eradication of H. pylori infection, substitution of ASA for other non-aspirin anti-platelet drugs, and co-therapy with misoprostol or H2RAs.

DETAILED DESCRIPTION:
No dose of "low-dose" aspirin (ASA) is safe in terms of the risk if ulcer bleeding. Even at a dose as low as 75 mg daily, ASA doubles the risk of ulcer bleeding when compared to the risk in non-users. This rise in the incidence was associated with a 44% increase in usage of ASA. In Hong Kong, ASA is also a major cause of peptic ulcer complications.

In the absence of safer aspirins, co-therapy with a gastroprotective drug remains the dominant preventive strategy. Given the vast number of people taking ASA, however, it is only cost-effective to identify and treat those who are at high risk of ulcer bleeding and who have a strong indication for ASA use. Data from observational studies and randomized trials have consistently shown that PPIs are effective in reducing the risk of ulcer bleeding associated with ASA. Other potential preventive strategies include eradication of H. pylori infection, substitution of ASA for other non-aspirin anti-platelet drugs, and co-therapy with misoprostol or H2RAs. Among these preventive strategies, co-therapy with a PPI for prevention of ulcer bleeding in high-risk ASA users remains the most studied and best proven strategy.

H2-receptor antagonists (H2RAs) are relatively weak acid suppressing drugs when compared to PPIs. Very few studies have evaluated the efficacy of H2RAs in the prevention of peptic ulcer bleeding with ASA. Two case-control studies yielded conflicting results with regard to the efficacy of H2RAs in reducing the risk of hospitalizations for ulcer bleeding with ASA. There is a limited data on the efficacy of H2RAs, however, our local health authority has endorsed the use of H2RA as a co-therapy in high-risk ASA users since 2001.

On the other hand, H2RAs have two potential advantages over PPIs. First, generic H2RAs are much cheaper than generic PPIs in Hong Kong. Second, unlike the interaction between PPIs and clopidogrel, concomitant use of H2RAs and clopidogrel is not associated with an increased risk of recurrent myocardial infarction. Thus, H2RA might be a cheap and safe gastroprotective drug in patients requiring dual anti-platelet therapy (i.e., ASA and clopidogrel) who require coronary stents.

In patients with acute coronary syndrome or acute ischemic stroke who develop ASA-induced bleeding peptic ulcers, whether ASA should be discontinued before ulcers have healed is a major dilemma. In another double-blind randomized trial, we have shown that discontinuation of ASA after endoscopic treatment of bleeding ulcers was associated with a significantly increased in mortality within 8 weeks.

The investigators aim to test the hypothesis that PPI is superior to H2RA for the prevention of recurrent upper gastrointestinal bleeding in ASA users with a history ulcer bleeding

ELIGIBILITY:
Inclusion Criteria:

1. A history of documented peptic ulcer bleeding (self-reported history without confirmation by the clinician is not acceptable)
2. Negative tests for H. pylori or successful eradication of H. pylori based on urease test or histology
3. Expected regular use of ASA for the duration of the trial
4. Age ≥ 18
5. Written informed consent obtained

Exclusion Criteria:

1. A history of gastric or duodenal surgery other than patch repair
2. Severe erosive esophagitis (LA grade C or D)
3. Gastric outlet obstruction
4. Terminal illness
5. Active malignancies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-01; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
recurrent non-variceal upper GI bleeding | 12 months
  defined as hematemesis, melena or a decrease in hemoglobin of at least 2 g/dL with ulcers or bleeding erosions confirmed by endoscopy, and adjudicated by an independent committee

SECONDARY OUTCOMES:
lower GI bleeding | 12 Months
  defined by either melena or rectal bleeding causing hospital admission or transfusion, with negative results on upper endoscopy, or by a decrease in hemoglobin of at least 2 g/dL in association with negative results on upper endoscopy and no other explanations for the anemia.
atherothrombotic events | 12 months
  atherothrombotic events
A composite of recurrent upper GI bleeding or recurrent endoscopic ulcers | 12 months
  defined as hematemesis, melena or a decrease in hemoglobin of at least 2 g/dL with ulcers or bleeding erosions confirmed by endoscopy, and adjudicated by an independent committee

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (8):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Japan (7):
  - Second Department of Internal Medicine, Shimane University Faculty of Medicine, Izumo, Japan, Izumo
  - Department of Molecular Gastroenterology and Hepatology, Kyoto Prefectural University of Medicine, Kyoto, Japan, Kyoto
  - Department of Gastroenterology, Osaka City General Hospital, Osaka, Japan (Satellite hospital of Osaka City University), Osaka
  - Department of Gastroenterology, Osaka City University Graduate School of Medicine, Osaka
  - Department of Gastroenterology, Takarazuka Municipal Hospital, Hyogo, Japan (Satellite hospital of Osaka City University), Osaka
  - Second Department of Internal Medicine, Osaka Medical College, Takatsuki, Osaka, Japan, Osaka
  - Department of Internal Medicine and Gastroenterology, Saga Medical School, Saga, Japan, Saga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan FK, Kyaw M, Tanigawa T, Higuchi K, Fujimoto K, Cheong PK, Lee V, Kinoshita Y, Naito Y, Watanabe T, Ching JY, Lam K, Lo A, Chan H, Lui R, Tang RS, Sakata Y, Tse YK, Takeuchi T, Handa O, Nebiki H, Wu JC, Abe T, Mishiro T, Ng SC, Arakawa T. Similar Efficacy of Proton-Pump Inhibitors vs H2-Receptor Antagonists in Reducing Risk of Upper Gastrointestinal Bleeding or Ulcers in High-Risk Users of Low-Dose Aspirin. Gastroenterology. 2017 Jan;152(1):105-110.e1. doi: 10.1053/j.gastro.2016.09.006. Epub 2016 Sep 15. PMID 27641510